CLINICAL TRIAL: NCT04445987
Title: A Phase 2, Multicenter, Open-Label Study of the Long-Term Safety of ARQ-154 Foam 0.3% in Subjects With Seborrheic Dermatitis
Brief Title: Long-Term Safety of ARQ-154 Foam in Subjects With Seborrheic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arcutis Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARQ-154-214
Record Dates: First submitted 2020-06-22; First posted 2020-06-24 (Actual); Results first posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-05

CONDITIONS: Seborrheic Dermatitis
MeSH Terms: conditions — Dermatitis, Seborrheic

STUDY DESIGN:
Intervention Model Description: Subjects that consent to enter this open-label safety study may or may not have previously completed a companion study (ARQ-154 trial)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Long-term safety of ARQ-154 (Experimental): Open-label, Long-term Safety of ARQ-154
  Interventions: Drug: ARQ-154

INTERVENTIONS:
Drug: ARQ-154 — ARQ-154 foam 0.3% applied once daily for 52 weeks

SUMMARY:
This is an open-label, long-term safety study of roflumilast ARQ-154 foam 0.3% in subjects with seborrheic dermatitis involving up to 20% total Body Surface Area (BSA). Study was applied topically once daily for 52 weeks. Cohort 1 subjects are rollover subjects from study ARQ-154-203 (NCT04091646) and were rolled into treatment in the current study without interruption. Cohort 2 includes participants from ARQ-154-203 who began treatment in the current study after a gap from completing treatment in the prior study.

ELIGIBILITY:
Inclusion Criteria:

1. Participants legally competent to sign and give informed consent or (for adolescents) assent.
2. Males and females ages 9 years and older (inclusive) at the time of consent.
3. Females of childbearing potential (FOCBP) must have a negative serum pregnancy test at all study visits.
4. Post-menopausal women with spontaneous amenorrhea for at least 12 months or have undergone surgical sterilization.

   Cohort 1 only:
5. Subjects with seborrheic dermatitis who met eligibility criteria for a prior ARQ-154 study, successfully completed a prior ARQ-154 study through final visit and are able to immediately enroll into this long-term safety study on the final visit of the previous ARQ-154 study.

   Cohort 2 subjects that have not participated in a prior ARQ-154 study:
6. Clinical diagnosis of seborrheic dermatitis of at least 3 months duration as determined by the Investigator. Stable disease for the past 4 weeks.
7. Seborrheic dermatitis of the scalp and/or face and/or trunk and/or intertriginous areas up to ≤20% BSA involvement.
8. An Investigator Global Assessment (IGA) of disease severity of at least Moderate ('3') at Day 1.
9. Overall Assessment of Erythema and Overall Assessment of Scaling scores of Moderate ('2') at Day 1.

   Cohort 2 subjects that have participated in a prior ARQ-154 study:
10. Clinical diagnosis of seborrheic dermatitis of at least 3 months duration as determined by the Investigator.
11. Seborrheic dermatitis of the scalp and/or face and/or trunk and/or intertriginous areas up to ≤20% BSA involvement.

Exclusion Criteria:

1. Planned excessive exposure of treated area(s) to either natural or artificial sunlight, tanning bed or other LED.
2. Subjects with any condition on the treatment area which, in the opinion of the Investigator, could confound efficacy measurements.
3. Subjects unable to apply investigational product to the scalp due to physical limitation.
4. Known allergies to excipients in ARQ-154 foam.
5. Subjects who cannot discontinue the use of strong P-450 cytochrome inhibitors e.g., indinavir, nelfinavir, ritonavir, clarithromycin, itraconazole, ketoconazole, nefazodone, saquinavir, suboxone and telithromycin during the study period.
6. Known or suspected:

   * severe renal insufficiency or moderate to severe hepatic disorders
   * history of severe depression, suicidal ideation or C-SSRS indicative of suicidal ideation, whether lifetime or recent/recurrent.
7. Females who are pregnant, wishing to become pregnant during the study, or are breast-feeding.
8. Subjects with any serious medical condition or laboratory abnormality that would prevent study participation or place the subject at significant risk, as determined by the Investigator.
9. Subjects with a history of chronic alcohol or drugs abuse within 6 months of initiation of investigational product.
10. Current or a history of cancer within 5 years with the exception of fully treated skin basal cell carcinoma, cutaneous squamous cell carcinoma or carcinoma in situ of the cervix.
11. Subjects who are unable to communicate, read or understand the local language, or who display another condition, which in the Investigator's opinion, makes them unsuitable for clinical study participation.
12. Subjects who are family members of the clinical study site, clinical study staff, or sponsor, or family members that live in the same household of enrolled subjects.

    Cohort 1 only:
13. Subjects who experienced an ARQ-154 treatment-related AE or a serious AE (SAE) that precluded further treatment with ARQ-154 foam in a prior ARQ-154 study.
14. Subjects that use any Excluded Medication and Treatments.

    Cohort 2 only:
15. Subjects who cannot discontinue treatment with therapies for the treatment of seborrheic dermatitis prior to the Day 1 visit and during the study according to Excluded Medications and Treatments.
16. Subjects with PHQ-8 >10 or modified PHQ-A >10 at Screening or Day 1.

    Cohort 2 subjects that have participated in a prior ARQ-154 study:
17. Subjects who experienced an ARQ-154 treatment-related AE or a serious AE (SAE) that precluded further treatment with ARQ-154 foam in a prior ARQ-154 study.

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 408 (Actual)
Dates: Start 2020-06-12 (Actual); Primary Completion 2022-11-19 (Actual); Study Completion 2022-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Berk, MD, Study Director — Arcutis Biotherapeutics
Locations (39):
- United States (39):
  - Arcutis Biotherapeutics Clinical Site 59, Beverly Hills, California
  - Arcutis Biotherapeutics Clinical Site 51, Encino, California
  - Arcutis Biotherapeutics Clinical Site 75, Fountain Valley, California
  - Arcutis Biotherapeutics Clinical Site 19, Fremont, California
  - Arcutis Biotherapeutics Clinical Site 62, Los Angeles, California
  - Arcutis Biotherapeutics Clinical Site 64, San Diego, California
  - Arcutis Biotherapeutics Clinical Site 21, Santa Monica, California
  - Arcutis Biotherapeutics Clinical Site 53, Aventura, Florida
  - Arcutis Biotherapeutics Clinical Site 42, Coral Gables, Florida
  - Arcutis Biotherapeutics Clinical Site 57, Delray Beach, Florida
  - Arcutis Biotherapeutics Clinical Site 24, Miami, Florida
  - Arcutis Biotherapeutics Clinical Site 65, Sanford, Florida
  - Arcutis Biotherapeutics Clinical Site 12, Tampa, Florida
  - Arcutis Biotherapeutics Clinical Site 10, Rolling Meadows, Illinois
  - Arcutis Biotherapeutics Clinical Site 22, Plainfield, Indiana
  - Arcutis Biotherapeutics Clinical Site 15, Louisville, Kentucky
  - Arcutis Biotherapeutics Clinical Site 52, Metairie, Louisiana
  - Arcutis Biotherapeutics Clinical Site 28, Rockville, Maryland
  - Arcutis Biotherapeutics Clinical Site 73, Brighton, Massachusetts
  - Arcutis Biotherapeutics Clinical Site 40, Clinton Township, Michigan
  - Arcutis Biotherapeutics Clinical Site 20, Detroit, Michigan
  - Arcutis Biotherapeutics Clinical Site 58, Fort Gratiot, Michigan
  - Arcutis Biotherapeutics Clinical Site 14, Fridley, Minnesota
  - Arcutis Biotherapeutics Clinical Site 50, Las Vegas, Nevada
  - Arcutis Biotherapeutics Clinical Site 56, Portsmouth, New Hampshire
  - Arcutis Biotherapeutics Clinical Site 55, New York, New York
  - Arcutis Biotherapeutics Clinical Site 63, The Bronx, New York
  - Arcutis Biotherapeutics Clinical Site 23, High Point, North Carolina
  - Arcutis Biotherapeutics Clinical Site 18, Bexley, Ohio
  - Arcutis Biotherapeutics Clinical Site 29, Portland, Oregon
  - Arcutis Biotherapeutics Clinical Site 27, Pittsburgh, Pennsylvania
  - Arcutis Biotherapeutics Clinical Site 76, Charleston, South Carolina
  - Arcutis Biotherapeutics Clinical Site 13, Arlington, Texas
  - Arcutis Biotherapeutics Clinical Site 11, Austin, Texas
  - Arcutis Biotherapeutics Clinical Site 41, College Station, Texas
  - Arcutis Biotherapeutics Clinical Site 25, Houston, Texas
  - Arcutis Biotherapeutics Clinical Site 26, Pflugerville, Texas
  - Arcutis Biotherapeutics Clinical Site 54, San Antonio, Texas
  - Arcutis Biotherapeutics Clinical Site 17, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alexis AF, Bukhalo M, Cook-Bolden FE, Del Rosso JQ, Draelos ZD, DuBois JC, Ferris LK, Forman SB, Kempers SE, Kircik LH, Lain E, Moore AY, Pariser DM, Raoof J, Zirwas MJ, Seal MS, Kato S, Chu DH, Krupa D, Snyder S, Burnett P, Berk DR. Long-Term Safety and Efficacy of Roflumilast Foam 0.3% in Patients with Seborrheic Dermatitis: A Phase II, Open-Label Trial of up to 52 Weeks. Am J Clin Dermatol. 2026 Jan;27(1):189-198. doi: 10.1007/s40257-025-00984-2. Epub 2025 Nov 1. PMID 41175336

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 39 study centers in the US.
Pre-assignment Details: Participants from study ARQ-154-203 were rolled over primarily into this study. A subset of participants from study ARQ-154-116 was also enrolled (Cohort 1 Group 2); these participants are not included in the efficacy analyses but baseline and safety information is presented.
Groups:
- Cohort 1 Group 1: ARQ-154-203 Roflumilast Foam 0.3% Without Treatment Gap: Participants from ARQ-154-203 using roflumilast (ARQ-154) foam 0.3% in the prior study applied roflumilast foam 0.3% QD for 52 weeks in the present study with no gap in treatment.
- Cohort 1 Group 1: ARQ 154-203 Vehicle Foam Rolled Over Without Treatment Gap: Participants from ARQ-154-203 using vehicle foam in the prior study applied roflumilast foam 0.3% QD for 52 weeks in the present study with no gap in treatment.
- Cohort 2 Group 3: ARQ-154-203 Roflumilast Foam 0.3% With Treatment Gap: Participants from ARQ-154-203 using roflumilast foam in the prior study applied roflumilast foam 0.3% QD for 52 weeks in the present study with a gap in treatment.
- Cohort 2 Group 3: ARQ-154-203 Vehicle Foam With Treatment Gap: Participants from ARQ-154-203 using vehicle foam in the prior study applied roflumilast foam 0.3% QD for 52 weeks in the present study with a gap in treatment.
- Cohort 2 Group 4: De Novo Participants: Treatment naive participants who had not previously participated in a clinical study of roflumilast foam 0.3% applied roflumilast foam 0.3% QD for 52 weeks in the present study.
- Cohort 1 Group 2: ARQ-154-116 Rollover: Participants from study ARQ-154-116 applied roflumilast foam 0.3% in the present study.
Period: Overall Study
Arm/Group | Cohort 1 Group 1: ARQ-154-203 Roflumilast Foam 0.3% Without Treatment Gap | Cohort 1 Group 1: ARQ 154-203 Vehicle Foam Rolled Over Without Treatment Gap | Cohort 2 Group 3: ARQ-154-203 Roflumilast Foam 0.3% With Treatment Gap | Cohort 2 Group 3: ARQ-154-203 Vehicle Foam With Treatment Gap | Cohort 2 Group 4: De Novo Participants | Cohort 1 Group 2: ARQ-154-116 Rollover
Started | 52 | 23 | 41 | 17 | 267 | 8
Completed | 43 | 20 | 37 | 16 | 211 | 7
Not Completed | 9 | 3 | 4 | 1 | 56 | 1
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 4 | 0
Not completed — Lost to Follow-up | 4 | 3 | 1 | 1 | 29 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 4 | 0 | 1 | 0 | 18 | 1
Not completed — Other reason | 0 | 0 | 1 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Efficacy data were not summarized for participants from Cohort 1 Group 2.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 Group 1: ARQ-154-203 Roflumilast Foam 0.3% Without Treatment Gap | Cohort 1 Group 1: ARQ 154-203 Vehicle Foam Rolled Over Without Treatment Gap | Cohort 2 Group 3: ARQ-154-203 Roflumilast Foam 0.3% With Treatment Gap | Cohort 2 Group 3: ARQ-154-203 Vehicle Foam With Treatment Gap | Cohort 2 Group 4: De Novo Participants | Cohort 1 Group 2: ARQ-154-116 Rollover | Total
Number analyzed (Participants) | 52 | 23 | 41 | 17 | 267 | 8 | 408
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.5 (15.99) | 41.0 (15.53) | 46.7 (17.20) | 48.8 (14.99) | 42.4 (16.45) | 13.5 (2.1) | 42.8 (16.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 9 | 21 | 8 | 138 | 4 | 207
  Male | 25 | 14 | 20 | 9 | 129 | 4 | 201
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 10 | 8 | 0 | 86 | 6 | 121
  Not Hispanic or Latino | 41 | 13 | 33 | 17 | 179 | 2 | 285
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 2 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 3 | 0 | 1 | 0 | 13 | 1 | 18
  Black or African-American | 5 | 2 | 4 | 2 | 38 | 0 | 51
  Native Hawaii or Other Pacific Islander | 0 | 0 | 0 | 0 | 1 | 0 | 1
  White | 42 | 19 | 36 | 15 | 207 | 6 | 325
  Other | 0 | 2 | 0 | 0 | 4 | 0 | 6
  More than one race | 2 | 0 | 0 | 0 | 1 | 1 | 4
  Missing | 0 | 0 | 0 | 0 | 3 | 0 | 3
Investigator Global Assessment (IGA) Baseline Score [Count of Participants; unit: Participants] — The IGA is a 5-point scale assessing the severity of seborrheic dermatitis, with scores ranging from 0 ('clear') to 4 ('severe'), and higher scores indicate greater symptom severity.
  Participants
    0 - Completely clear | 0 | 2 | 0 | 0 | 0 | 0 | 2
    1 = Almost clear | 0 | 7 | 0 | 2 | 0 | 0 | 9
    2 = Mild | 0 | 2 | 0 | 2 | 0 | 0 | 4
    3 = Moderate | 44 | 11 | 38 | 13 | 235 | 5 | 346
    4 = Severe | 8 | 1 | 3 | 0 | 32 | 3 | 47

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With ≥1 Adverse Event (AE)
Description: The number of participants with treatment-emergent AEs is reported. An AE is any untoward or unfavorable medical occurrence in a human participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to participation in the research. Data are presented according to cohort group assigned as treatment were identical in this study regardless of the treatment received in the prior study.
Time Frame: Up to 52 weeks
Population: All participants are included.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1 Group 1: ARQ-154-203 Roflumilast Foam 0.3% Without Treatment Gap: Participants from ARQ-154-203 using either roflumilast foam 0.3% or vehicle foam in the prior study applied roflumilast foam 0.3% QD for 52 weeks in the present study with no gap in treatment.
- Cohort 2 Groups 3 and 4: ARQ-154-203 Roflumilast Foam 0.3% With Treatment Gap: Participants from ARQ-154-203 using roflumilast foam 0.3% or vehicle foam in the prior study applied roflumilast foam 0.3% QD for 52 weeks in the present study with a gap in treatment.
Arm/Group | Cohort 1 Group 1: ARQ-154-203 Roflumilast Foam 0.3% Without Treatment Gap | Cohort 2 Groups 3 and 4: ARQ-154-203 Roflumilast Foam 0.3% With Treatment Gap | Cohort 2 Group 4: De Novo Participants | Cohort 1 Group 2: ARQ-154-116 Rollover
Number analyzed (Participants) | 75 | 58 | 267 | 8
Participants | 17 | 23 | 90 | 3

2. Primary Outcome: Number of Participants With ≥1 Serious Adverse Event (SAE)
Description: The number of participants with treatment-emergent SAEs is reported. An SAE is any AE that results in death, is life-threatening (places the subject at immediate risk of death from the event as it occurred), requires inpatient hospitalization or prolongation of existing hospitalization, results in a persistent or significant disability/incapacity, results in a congenital anomaly/birth defect, or is any other adverse event that, based upon appropriate medical judgment, may jeopardize the subject's health. Data are presented according to cohort group assigned as treatment were identical in this study regardless of the treatment received in the prior study.
Time Frame: Up to 52 weeks
Population: All participants are included.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1 Group 1: ARQ-154-203 Roflumilast Foam 0.3% Without Treatment Gap: Participants from ARQ-154-203 using roflumilast (ARQ-154) foam 0.3% or vehicle foam in the prior study applied roflumilast foam 0.3% QD for 52 weeks in the present study with no gap in treatment.
- Cohort 2 Group 3: ARQ-154-203 Roflumilast Foam 0.3% With Treatment Gap: Participants from ARQ-154-203 using vehicle foam in the prior study applied roflumilast foam 0.3% QD for 52 weeks in the present study with a gap in treatment.
Arm/Group | Cohort 1 Group 1: ARQ-154-203 Roflumilast Foam 0.3% Without Treatment Gap | Cohort 2 Group 3: ARQ-154-203 Roflumilast Foam 0.3% With Treatment Gap | Cohort 2 Group 4: De Novo Participants | Cohort 1 Group 2: ARQ-154-116 Rollover
Number analyzed (Participants) | 75 | 58 | 267 | 8
Participants | 2 | 0 | 5 | 0

3. Secondary Outcome: Number of Participants With an Investigator Global Assessment (IGA) Score of Completely Clear or Almost Clear
Description: The number of participants with an IGA score of 0 ('completely clear') or 1 ('almost clear') is presented. The IGA is a 5-point scale assessing the severity of seborrheic dermatitis, with scores ranging from 0 ('clear') to 4 ('severe'), and higher scores indicate greater symptom severity.
Time Frame: Weeks 4, 12, 24, 36, and 52
Population: All treated participants with data available and who had baseline IGA score >1 are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 Group 1: ARQ-154-203 Roflumilast Foam 0.3% Without Treatment Gap | Cohort 1 Group 1: ARQ 154-203 Vehicle Foam Rolled Over Without Treatment Gap | Cohort 2 Group 3: ARQ-154-203 Roflumilast Foam 0.3% With Treatment Gap | Cohort 2 Group 3: ARQ-154-203 Vehicle Foam With Treatment Gap | Cohort 2 Group 4: De Novo Participants | Cohort 1 Group 2: ARQ-154-116 Rollover
Number analyzed (Participants) | 52 | 23 | 41 | 17 | 267 | 7
Participants
  Week 4: number analyzed (Participants) | 50 | 13 | 39 | 15 | 260 | 7
  Week 4 | 36 | 7 | 20 | 10 | 137 | 5
  Week 12: number analyzed (Participants) | 47 | 13 | 38 | 15 | 242 | 7
  Week 12 | 35 | 7 | 25 | 12 | 172 | 5
  Week 24: number analyzed (Participants) | 44 | 12 | 37 | 14 | 225 | 3
  Week 24 | 31 | 10 | 24 | 11 | 177 | 3
  Week 36: number analyzed (Participants) | 0 | 0 | 1 | 2 | 47 | 0
  Week 36 |  |  | 0 | 0 | 37 |
  Week 52: number analyzed (Participants) | 0 | 0 | 1 | 1 | 43 | 0
  Week 52 |  |  | 1 | 1 | 35 |

4. Secondary Outcome: Achievement of IGA Success
Description: The number of participants achieving "success" in IGA assessment of disease severity is presented. Success was defined as achievement of an IGA score of 0 ('clear') or 1 ('almost clear') at Week 8, accompanied by a ≥2-grade improvement from baseline IGA score. The IGA is a 5-point scale assessing the severity of seborrheic dermatitis, with scores ranging from 0 ('clear') to 4 ('severe'), and higher scores indicate greater symptom severity.
Time Frame: Weeks 4, 12, 24, 36, and 52
Population: All treated participants with data available and who had baseline IGA score ≥2 are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 Group 1: ARQ-154-203 Roflumilast Foam 0.3% Without Treatment Gap | Cohort 1 Group 1: ARQ 154-203 Vehicle Foam Rolled Over Without Treatment Gap | Cohort 2 Group 3: ARQ-154-203 Roflumilast Foam 0.3% With Treatment Gap | Cohort 2 Group 3: ARQ-154-203 Vehicle Foam With Treatment Gap | Cohort 2 Group 4: De Novo Participants | Cohort 1 Group 2: ARQ-154-116 Rollover
Number analyzed (Participants) | 50 | 22 | 39 | 17 | 260 | 7
Participants
  Week 4: number analyzed (Participants) | 50 | 13 | 39 | 15 | 260 | 7
  Week 4 | 36 | 6 | 20 | 8 | 137 | 5
  Week 12: number analyzed (Participants) | 47 | 13 | 38 | 15 | 242 | 7
  Week 12 | 35 | 7 | 25 | 11 | 172 | 5
  Week 24: number analyzed (Participants) | 44 | 12 | 37 | 14 | 225 | 3
  Week 24 | 31 | 10 | 24 | 11 | 177 | 3
  Week 36: number analyzed (Participants) | 0 | 0 | 1 | 1 | 47 | 0
  Week 36 | 0 | 0 | 0 | 0 | 37 | 0
  Week 52: number analyzed (Participants) | 0 | 0 | 1 | 1 | 43 | 0
  Week 52 | 0 | 0 | 1 | 1 | 35 | 0

5. Secondary Outcome: Duration of IGA Success
Description: The duration of "success" in IGA assessment of disease severity is presented. Success was defined as achievement of an IGA score of 0 ('clear') or 1 ('almost clear') at Week 8, accompanied by a ≥2-grade improvement from baseline IGA score. The IGA is a 5-point scale assessing the severity of seborrheic dermatitis, with scores ranging from 0 ('clear') to 4 ('severe'), and higher scores indicate greater symptom severity. The time from first observation of IGA success to the first subsequent time a participant's disease response did not meet the criteria for IGA success is presented. The duration of IGA success for subjects who ended treatment in IGA success was censored at the last disease assessment date.
Time Frame: Weeks 4, 12, 24, 36, and 52
Population: All treated participants who achieved IGA success and had data available are included.
Measure: Median (Full Range); unit: weeks
Arm/Group | Cohort 1 Group 1: ARQ-154-203 Roflumilast Foam 0.3% Without Treatment Gap | Cohort 1 Group 1: ARQ 154-203 Vehicle Foam Rolled Over Without Treatment Gap | Cohort 2 Group 3: ARQ-154-203 Roflumilast Foam 0.3% With Treatment Gap | Cohort 2 Group 3: ARQ-154-203 Vehicle Foam With Treatment Gap | Cohort 2 Group 4: De Novo Participants | Cohort 1 Group 2: ARQ-154-116 Rollover
Number analyzed (Participants) | 50 | 11 | 61 | 35 | 229 | 6
weeks | 18.786 [0.14 to 32.29] | 12.143 [0.14 to 22.29] | 7.714 [0.14 to 30.43] | 13.143 [0.14 to 31.86] | 19.00 [0.14 to 50.14] | 10.00 [3.57 to 23.71]

6. Secondary Outcome: IGA Treatment-Free Interval
Description: The treatment-free interval is defined as time from when the participant achieves disease clearance (IGA score of 0 ["completely clear"]) and stops treatment of all lesions until the time of restarting treatment.
Time Frame: Weeks 4, 12, 24, 36, and 52
Population: All treated participants who achieved an IGA score of 0 are included.
Measure: Median (Full Range); unit: weeks
Arm/Group | Cohort 1 Group 1: ARQ-154-203 Roflumilast Foam 0.3% Without Treatment Gap | Cohort 1 Group 1: ARQ 154-203 Vehicle Foam Rolled Over Without Treatment Gap | Cohort 2 Group 3: ARQ-154-203 Roflumilast Foam 0.3% With Treatment Gap | Cohort 2 Group 3: ARQ-154-203 Vehicle Foam With Treatment Gap | Cohort 2 Group 4: De Novo Participants | Cohort 1 Group 2: ARQ-154-116 Rollover
Number analyzed (Participants) | 15 | 8 | 18 | 7 | 90 | 3
weeks | 19.143 [0.57 to 24.00] | 11.766 [2.57 to 24.43] | 11.929 [1.14 to 22.14] | 14.143 [2.43 to 22.00] | 12.143 [0.29 to 49.14] | 20.143 [8.143 to 23.14]

ADVERSE EVENTS:
Time Frame: Up to 52 weeks
Description: All participants are included. Data are presented according to cohort group assigned as treatment were identical in this study regardless of the treatment received in the prior study.
Groups:
- Cohort 1 Group 1: ARQ-154-203 Roflumilast Foam 0.3% Without Treatment Gap: Participants from ARQ-154-203 using roflumilast foam 0.3% or vehicle foam in the prior study applied roflumilast foam 0.3% QD for 52 weeks in the present study with no gap in treatment.
- Cohort 2 Group 3: ARQ-154-203 Roflumilast Foam 0.3% Without Treatment Gap: Participants from ARQ-154-203 using roflumilast 0.3% or vehicle foam in the prior study applied roflumilast foam 0.3% QD for 52 weeks in the present study with a gap in treatment.
Arm/Group | Cohort 1 Group 1: ARQ-154-203 Roflumilast Foam 0.3% Without Treatment Gap | Cohort 2 Group 3: ARQ-154-203 Roflumilast Foam 0.3% Without Treatment Gap | Cohort 2 Group 4: De Novo Participants | Cohort 1 Group 2: ARQ-154-116 Rollover
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/58 | 1/267 | 0/8
Serious Adverse Events (participants affected / at risk) | 2/75 | 0/58 | 5/267 | 0/8
Other Adverse Events (participants affected / at risk) | 3/75 | 4/58 | 11/267 | 6/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 Group 1: ARQ-154-203 Roflumilast Foam 0.3% Without Treatment Gap (N=75) | Cohort 2 Group 3: ARQ-154-203 Roflumilast Foam 0.3% Without Treatment Gap (N=58) | Cohort 2 Group 4: De Novo Participants (N=267) | Cohort 1 Group 2: ARQ-154-116 Rollover (N=8)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Performance status decreased (General disorders) | 0 | 0 | 1 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 Group 1: ARQ-154-203 Roflumilast Foam 0.3% Without Treatment Gap (N=75) | Cohort 2 Group 3: ARQ-154-203 Roflumilast Foam 0.3% Without Treatment Gap (N=58) | Cohort 2 Group 4: De Novo Participants (N=267) | Cohort 1 Group 2: ARQ-154-116 Rollover (N=8)
COVID-19 (Infections and infestations) | 3 | 3 | 9 | 0
Urinary tract infection (Infections and infestations) | 0 | 4 | 3 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 1
Tic (Psychiatric disorders) | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Application site alopecia (General disorders) | 0 | 0 | 0 | 1
Transaminases increased (Investigations) | 0 | 0 | 0 | 1
Pyogenic granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor is supportive of publishing clinical trial findings. The process of coordinating publication efforts is detailed in the Clinical Trial Agreement.

DOCUMENTS (2):
  • Study Protocol (2021-11-04): https://cdn.clinicaltrials.gov/large-docs/87/NCT04445987/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-18): https://cdn.clinicaltrials.gov/large-docs/87/NCT04445987/SAP_001.pdf